CLINICAL TRIAL: NCT04122079
Title: Validation of the Spanish Version of the Clinical Outcomes in Routine Evaluation-Outcome Measure (CORE-OM) in Chile
Status: Completed | Type: Observational
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Other Study IDs: 181130009
Record Dates: First submitted 2019-10-02; First posted 2019-10-10 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2019-10

CONDITIONS: Psychological Distress
Keywords: CORE-OM; Outcome measures; Psychometric validation; Psychological distress

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Clinical (outpatients): Patients receiving mental health treatment at the three psychotherapeutic centers; two university clinics and a family mental health clinic
- Clinical (self-reported): Students and community nonstudent participants who were receiving psychological or psychiatric treatment
- Non-clinical (Community): Members of the community
- Non-clinical (Students): University undergraduate students

SUMMARY:
AIM: study the psychometric properties of the Spanish version of the Clinical Outcomes in Routine Evaluation-Outcome Measure (CORE-OM), an instrument that measures psychological distress, in the Chilean population.

SAMPLES: two clinical samples (1. outpatients from three psychotherapeutic centers; two university clinics and a family mental health clinic and 2. self-reported clinical) and two non-clinical (1. university students; and 2. general community) samples. Students and community nonstudent participants who reported receiving psychological or psychiatric treatment (exclusion criterion) were excluded from the non-clinical sample and classified as self-reported clinical.

DATA COLLECTION: In the clinical sample, data (paper questionnaire) is collected at one point if the patient is undergoing treatment and at four points (at baseline (i.e. before the first session), at 2, 5 and 8-weeks) if the patient is recruited before attending the first psychotherapy session. Participants from the second university outpatient clinic and a family mental health clinic complete a digital version. At baseline, participants are presented with the CORE-OM and the Outcome Questionnaire (OQ-45). At each follow-up point, they are presented with the CORE-OM plus mental health service evaluation items.

In the student and community samples, data is collected at two time points (i.e. baseline and retest). At baseline, participants are presented with the CORE-OM and OQ-45. After two weeks (i.e. retest) participants are presented with the CORE-OM.

The application modality in the non-clinical samples is mixed: students and general community participants complete paper or digital versions of the questionnaire in the classroom or community, respectively.

RECRUITMENT: The clinical sample is recruited at two university outpatient clinics and a family mental health clinic of Santiago.

The student sample is recruited in classrooms. The general community sample is recruited using a convenience sampling method. As in other samples, participants sign an informed consent before answering the questionnaire.

ANALYSES: internal consistency, test-retest stability, convergent validity and discrimination. Clinical cut-off values will be calculated by domain and sex between the clinical and non-clinical samples and sensitivity to change will be assessed using data from the subsample of outpatients who respond an online questionnaire before their first session and at one follow up point.

DETAILED DESCRIPTION:
The AIM is to study the psychometric properties of the Spanish version of the Clinical Outcomes in Routine Evaluation-Outcome Measure (CORE-OM), an instrument that measures psychological distress, in the Chilean population.

To test internal consistency, test-retest stability, convergent validity and discrimination, the CORE-OM is applied in four SAMPLES: two clinical samples (1. outpatients from three psychotherapeutic centers; two university clinics and a family mental health clinic (n=200 ~) and 2. self-reported clinical (n=200 ~)) and two non-clinical (1. university students (n=400 ~); and 2. general community (n=300~)) samples. Students and community nonstudent participants who reported receiving psychological or psychiatric treatment (exclusion criterion) were excluded from the non-clinical sample and classified as self-reported clinical.

Specific modalities of DATA COLLECTION are used for each sample. In the clinical sample, data is collected at one time point if the patient is undergoing treatment and at four time points (at baseline (i.e. before the first session), at 2 weeks (follow-up 1), at 5 weeks (follow-up 2), and at 8 weeks (follow-up 3)) if the patient is recruited before attending the first session of psychotherapy. Participants in the clinical sample complete a paper version of the questionnaire in the waiting room of one of the university outpatient clinics. Participants from the second university outpatient and family mental health clinics complete a digital version programmed in Google forms. At baseline, participants are presented with the CORE-OM, the Outcome Questionnaire (OQ-45) and a set of sociodemographic and mental health service use items. At each follow-up point they are presented with the CORE-OM plus mental health service evaluation items.

In the student and community samples, data is collected at two time points (i.e. baseline and retest). At baseline, participants are presented with the CORE-OM, OQ-45 and a set of sociodemographic and mental health service use items. After two weeks (i.e. retest) participants are presented with the CORE-OM plus an item about mental health service use in the last 30 days.

Student and community participants are contacted via email after 2 weeks to respond the online retest questionnaire.

The application modality in the non-clinical samples is mixed: students and general community participants complete paper or digital versions of the questionnaire in the classroom or community, respectively. The digital version of the questionnaire is in surveygizmo™ and can be accessed by clicking a Uniform Resource Locator (URL) embedded in an email/message, or by scanning a Quick Response (QR) code with a smartphone.

RECRUITMENT: The clinical sample is recruited at two university outpatient clinics and a family mental health clinic of Santiago, Chile all of which provide services to patients of low to medium income. Patients in one of the university clinics are approached by research assistants in the waiting area, before or after their psychotherapy/psychiatry session. Patients meeting inclusion criteria, and willing to participate, fill out an informed consent before responding the questionnaire. Patients form the second university clinic and the family mental health clinic are referred when booking their first appointment and contacted via email by a member of the research team. Questionnaire completion and responses to risk items are reviewed within 24 hours. Treating psychiatrists/psychologists are contacted via email when their patients respond "often" or "most of the time" to items signaling self-harm and thoughts of suicide (i.e. items 9, 16, 24 and 34 of the CORE-OM or item 8 of the OQ-45).

The student sample is recruited in the classrooms of Pontificia Universidad Católica de Chile. A member of the research team presents the study and invites students to participate. Students agreeing to participate fill out an informed consent form before completing paper/digital versions of the questionnaire. Any student responding "often" or "most of the time" to items signaling self-harm and thoughts of suicide in the CORE-OM/OQ-45 receives an email from the Responsible Investigator with information about the University´s counseling services within 24 hours.

The general community sample is recruited using a convenience sampling method (e.g. contacts of research team). As in the other samples, participants sign an informed consent before answering the questionnaire.

Since the non-clinical samples serve to test stability, students/general community are asked to provide a valid email address in order to send them an email invitation after two weeks to complete the CORE-OM.

Clinical cut-off values will be calculated by domain and sex between the clinical and non-clinical samples and sensitivity to change will be assessed using data from the subsample of outpatients who respond an online questionnaire before their first session and at one follow up point.

ELIGIBILITY:
Inclusion Criteria:

* Born in Chile
* Currently receiving mental health treatment at the University Outpatient Clinic (Centro Médico San Joaquín) (only Clinical Sample)
* Currently enrolled at the Universidad Catolica de Chile (only Student Sample)

Exclusion Criteria:

* Aged < 18
* Currently receiving psychological, psychiatric or neurological treatment (only Student and Community Sample)
* Full-time students (only Community Sample)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Four samples:
  1. Clinical (outpatients)
  2. Clinical (self-reported patients): university students or non-student community participant who report receiving mental health treatment
  2. Non-clinical (University students) 3. Non-clinical (Community)
Sampling Method: Non-Probability Sample
Enrollment: 1120 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Clinical Outcomes in Routine Evaluation Outcome Measure (CORE-OM). | Baseline
  A self-report questionnaire which measures general psychological distress
  It consists of 34 items that assess four domains:
  1. Well-being (W)
  2. Problems/Symptoms (P)
  3. Functioning (F)
  4. Risk (R)
  Each of the 34 items is scored on a 5-point scale ranging from 0 to 4. A total psychological distress score, ranging from 0 to136, can be calculated by adding all items, with higher scores indicating higher levels of psychological distress. A Well-Being dimension score, ranging from 0 to 16, can be calculated with higher scores indicating lower levels of subjective wellbeing. A Problems/Symptoms dimension score, ranging from 0 to 48, can be calculated with higher scores indicating higher levels of reported problems/distress. A Functioning dimension score, ranging from 0 to 48, can be calculated with higher scores indicating lower levels of functioning. A Risk dimension score, ranging from 0 to 24, can be calculated with higher scores indicating a greater level of risk.
Change from baseline on the Clinical Outcomes in Routine Evaluation Outcome Measure (CORE-OM) at 2 to 3 weeks. | Follow-up after two to three weeks (non-clinical sample)
  A self-report questionnaire which measures general psychological distress
  It consists of 34 items that assess four domains:
  1. Well-being (W)
  2. Problems/Symptoms (P)
  3. Functioning (F)
  4. Risk (R)
  Each of the 34 items is scored on a 5-point scale ranging from 0 to 4. A total psychological distress score, ranging from 0 to136, can be calculated by adding all items, with higher scores indicating higher levels of psychological distress. A Well-Being dimension score, ranging from 0 to 16, can be calculated with higher scores indicating lower levels of subjective wellbeing. A Problems/Symptoms dimension score, ranging from 0 to 48, can be calculated with higher scores indicating higher levels of reported problems/distress. A Functioning dimension score, ranging from 0 to 48, can be calculated with higher scores indicating lower levels of functioning. A Risk dimension score, ranging from 0 to 24, can be calculated with higher scores indicating a greater level of risk.
Change from baseline on the Clinical Outcomes in Routine Evaluation Outcome Measure (CORE-OM) at 2 to 3 weeks. | Follow-up after two, five and eight weeks (clinical sample)
  A self-report questionnaire which measures general psychological distress
  It consists of 34 items that assess four domains:
  1. Well-being (W)
  2. Problems/Symptoms (P)
  3. Functioning (F)
  4. Risk (R)
  Each of the 34 items is scored on a 5-point scale ranging from 0 to 4. A total psychological distress score, ranging from 0 to136, can be calculated by adding all items, with higher scores indicating higher levels of psychological distress. A Well-Being dimension score, ranging from 0 to 16, can be calculated with higher scores indicating lower levels of subjective wellbeing. A Problems/Symptoms dimension score, ranging from 0 to 48, can be calculated with higher scores indicating higher levels of reported problems/distress. A Functioning dimension score, ranging from 0 to 48, can be calculated with higher scores indicating lower levels of functioning. A Risk dimension score, ranging from 0 to 24, can be calculated with higher scores indicating a greater level of risk.
Outcome Questionnaire (OQ45/OQ45.2) | Baseline
  A self-report questionnaire which measures general psychological distress and is designed to monitor treatment outcomes in mental health settings.
  It consists of 45 items and contains three subscales:
  1. Symptom Distress (SD)
  2. Interpersonal Relations (IR)
  3. Social Role (SR)
  The OQ-45 provides a total score, ranging from 0 to 180, and three subscores per subscale. Symptom Distress (SD) scores range from 0 to 100, Interpersonal Relations (IR) scores range from 0 to 44 and Social Role (SR) scores range from 0 to 36.
  Higher scores reflect increased psychological distress associateed to experiencing a high number of symptoms (SD), interpersonal difficulties (IR), and/or decreased satisfaction and quality of life (SR). The clinical cut-off scores in the Chilean population are: SD=43; IR=16; SR=14 and Total Score=73.

CONTACTS AND LOCATIONS:
Overall Officials: Antonia Errazuriz, PhD, Principal Investigator — Universidad Catolica de Chile
Locations (1):
- Pontificia Universidad Catolica de Chile, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: Yes
IPD and related data dictionaries is available to researchers via Dataverse
Supporting Information: SAP, ICF
Time Frame: Currently available
Access Criteria: For research use (authorization by PI)
URL: https://doi.org/10.7910/DVN/IPNZYR

REFERENCES:
- [Background] Evans, C., Mellor-Clark, J., Margison, F., Barkham, M., Audin, K., Connell, J., & McGrath, G. (2000). CORE: Clinical Outcomes in Routine Evaluation. Journal of Mental Health, 9(3), 247-255
- [Background] Evans C, Connell J, Barkham M, Margison F, McGrath G, Mellor-Clark J, Audin K. Towards a standardised brief outcome measure: psychometric properties and utility of the CORE-OM. Br J Psychiatry. 2002 Jan;180:51-60. doi: 10.1192/bjp.180.1.51. PMID 11772852
- [Background] Von Bergen A., De la Parra G. (2002). OQ-45.2, Cuestionario para la evaluación de resultados y evolución en psicoterapia: adaptación, validación e indicaciones para su aplicación e interpretación [Questionnaire for the evaluation of results and evolution in psychotherapy: adaptation, validation and indications for its application and interpretation]. Ter. Psicol. 20 161-176
- [Result] Errazuriz A, Passi Solar A, Beltran R, Paz C, Evans C, De la Parra G. Psychometric properties of the Spanish version of the Clinical Outcomes in Routine Evaluation Outcome Measure (CORE-OM) in Chile. Psychother Res. 2025 Jul;35(6):1017-1029. doi: 10.1080/10503307.2024.2356195. Epub 2024 May 23. PMID 38781596